CLINICAL TRIAL: NCT03211052
Title: A Randomised Phase II Study of Neoadjuvant TAK-700 and Leuprorelin Acetate Followed by Surgery Versus Surgery Alone in Intermediate and High Risk Clinically Localized Prostate Cancer
Brief Title: A Study of Neoadjuvant TAK-700 and Leuprorelin Acetate Followed by Surgery Versus Surgery Alone
Acronym: NEPTUNE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IMP no longer available
Sponsor: Centre of Experimental Medicine (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Centre of Experimental Medicine, Professor Thomas Powles, Queen Mary University of London
Organization: Queen Mary University of London (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 008285QM
Record Dates: First submitted 2013-04-26; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel; Gonadotropin-Releasing Hormone; Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAK-700 + LHRH agonist + Prostatectomy (Experimental): Neoadjuvant TAK-700 for 6 months with LHRH agonists prior to prostatectomy
  Interventions: Drug: TAK-700 and LHRH agonist
- Prostatectomy (Other): Prostatectomy only-Within 28 days of randomisation
  Interventions: Procedure: prostatectomy

INTERVENTIONS:
Drug: TAK-700 and LHRH agonist — TAK-700 for 6 months 300mg BD with Leuprorelin Acetate Injections prior to planned prostatectomy
  Other Names: Orteronel (TAK 700); LHRH-Leuprorelin Acetate
  Arms: TAK-700 + LHRH agonist + Prostatectomy
Procedure: prostatectomy — SURGICAL REMOVAL OF THE PROSTATE
  Arms: Prostatectomy

SUMMARY:
This study investigates neoadjuvant TAK-700 orteronel for 6 months prior to prostatectomy. The three year biochemical free survival is the primary endpoint. There are a number of 2nd endpoints such as pathological complete response rate, the need for adjuvant radiation therapy, use of post operative radiotherapy an the rate of positive margins at surgery. Translational endpoints include measuring tumoural and plasma testosterone as well as other androgens.

Patients with untreated high risk and intermediate risk operable prostate cancer will be treated with TAK-700 (plus LHRH agonist) for 24 weeks prior to planned prostatectomy.

DETAILED DESCRIPTION:
Study Objectives:

To investigate if neoadjuvant TAK-700 with LHRH agonists and prostatectomy is associated with a delay in progression free survival compared to prostatectomy alone

To evaluate response (CR and PR) after at least 12 and 24 weeks of treatment with the study drugs Collection of Plasma, tissue and functional imaging with MRI To evaluate (molecular) expression of AR regulated genes and tumour immunohistochemistry. Molecular and protein expression will be correlated with intracellular androgen levels and pathologic response to ADT

136 patients will be randomised to this study. 68 patients will receive neoadjuvant therapy with TAK-700 and Leuprorelin Acetate followed by surgery and 68 patients will receive surgery alone.

This trial aims to recruit 136 patients with clinically localised prostate cancer. Patients will be stratified according to National Comprehensive Cancer Network (NCCN) risk stratification criteria and type of planned surgery. Definitions of risk categories can be found in the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. No previous treatment for prostate cancer (including surgery, any hormone therapy, radiotherapy, cryotherapy).
3. Age ≥ 18 years and male
4. Histologically or cytologically confirmed adenocarcinoma of the prostate with Gleason score. A prostate biopsy within 6 months from screening is allowed for entry requirements.
5. Intermediate or high risk prostate cancer according to National Comprehensive Cancer Network (NCCN) risk stratification criteria

   * Intermediate: PSA >10 & <20 or a Gleason score 7 or clinical stage up to and including T2c disease
   * High risk: PSA>20 or Gleason 8-10 or clinical stage >T2c
6. Serum testosterone > 200 ng/dL
7. Prostatectomy is the planned treatment option.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
9. Adequate organ function, defined as follows:

   * Hemoglobin >10.0g/dL
   * Absolute neutrophil count > 1.5 x 10.9/L
   * Platelet count >100 x 10.9/L
   * AST and /or ALT <2.5 x ULN
   * Total Bilirubin <1.5 x ULN

Exclusion Criteria:

1. Serious co-existent medical conditions such as chronic active autoimmune disease, (within the last 6 months) or infection (such as hepatitis).
2. Uncontrolled hypertension within the screening period (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg). Patients with a history of hypertension are allowed to enrol provided blood pressure is controlled by anti-hypertensive therapy.
3. Patients taking regular oral steroids for any reason.
4. Previously treated prostate cancer (including radiotherapy, hormone therapy or surgery).
5. History of pituitary or adrenal dysfunction
6. Other active malignancy over the last 5 years that has required systemic therapy excluding:

   1. Adjuvant therapy in the curative setting
   2. Non-melanoma skin cancer
   3. Superficial transitional cell carcinoma (CIS-T1).
7. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
8. Current enrolment in an investigational drug or device study or participation in such a study within 30 days of Day 1
9. Not willing to comply with the procedural requirements of this protocol, including repeat prostate biopsies
10. Patients who have partners of childbearing potential who are not willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 16 weeks after last study drug administration.
11. Uncontrolled diabetes mellitus, in the opinion of the treating physician
12. Known hypersensitivity to compounds related to TAK-700 or to TAK-700 excipients.
13. Hypersensitivity to any of the ingredients or to synthetic Gn-RH or Gn-RH derivatives.
14. Screening calculated ejection fraction of <50% by echocardiogram.
15. History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 (NCI CTCAE, version 4.02), thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (e.g., pericardial effusion restrictive cardiomyopathy) within 6 months prior to first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
16. New York Heart Association Class III or IV heart failure
17. ECG abnormalities of Q-wave infarction, unless identified 6 or more months prior to screening
18. QTc interval > 460 msec on ECG

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-06-02 (Actual)

PRIMARY OUTCOMES:
3 year biochemical progression free survival (PSA) | 3 years
  Post-operative serum PSA of greater or equal to 0.2 ng/dl on 2 separate occasions as defined by the AUA.

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom